CLINICAL TRIAL: NCT00579761
Title: A Retrospective Review of the Management of Infective Endocarditis in Patients at Virginia Commonwealth University Medical Center From 1996-2006
Brief Title: Retrospective Review of Management of Infective Endocarditis
Status: Withdrawn | Type: Observational
Why Stopped: Per PI on 12/9/15 - No patients were ever enrolled in this study
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM10420
Record Dates: First submitted 2007-12-17; First posted 2007-12-24 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Endocarditis
Keywords: Endocarditis; neurological deficit
MeSH Terms: conditions — Endocarditis; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an analysis of the outcomes of patients having undergone surgical intervention for infective endocarditis.

DETAILED DESCRIPTION:
This study will look at the presentations, epidemiology, risk factors, modalities of diagnosis; and the role of specific investigatory tools with surgical intervention and timimg of intervention in patients who underwent surgical treatment for infective endocarditis. Morbidity and Mortality post surgery and prognosis including long term outcome of our patients will be analyzed. Special attention will be made to those patients with pre-operative neurological deficit.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone surgical treatment for infective endocarditis

Exclusion Criteria:

* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects that have undergone surgical treatment for infective endocarditis at VCU medical Center from 1996 to present
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vigneshwar Kasirajan, MD, Principal Investigator — Virginia Commonwealth University Department of Cardiothoracic Surgery
Locations (1):
- Virginia Commonweath University MCV Hospital, Richmond, Virginia, United States